CLINICAL TRIAL: NCT01964872
Title: A Double Blind, Placebo-Controlled, Randomized, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-38877618 in Healthy Male Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ-38877618 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR102784; 38877618EDI1001 (Other: Janssen Cilag N.V./S.A., Belgium); 2013-002551-16 (EudraCT Number)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; JNJ-38877618; Pharmacokinetic; Safety; Single-ascending dose; Multiple-ascending dose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-38877618 (Experimental)
  Interventions: Drug: JNJ-38877618: Part 1a; Drug: JNJ-38877618: Part 1b; Drug: JNJ-38877618: Part 1c (optional); Drug: JNJ-38877618: Part 2; Drug: JNJ-38877618: Part 3; Drug: JNJ-38877618: Part 4 (optional)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo: Parts 1a, 2, 3, and 4 (optional)

INTERVENTIONS:
Drug: JNJ-38877618: Part 1a — Single ascending dose administered orally in liquid formulation (Formulation A). The planned dose range for Parts 1 and 2 will be 6 to 1200 mg.
  Arms: JNJ-38877618
Drug: JNJ-38877618: Part 1b — Single dose administered orally in capsule formulation (Formulation B). The planned dose range for Parts 1 and 2 will be 6 to 1200 mg.
  Arms: JNJ-38877618
Drug: JNJ-38877618: Part 1c (optional) — Single dose administered orally in an alternative capsule formulation (Formulation C). The planned dose range for Parts 1 and 2 will be 6 to 1200 mg.
  Arms: JNJ-38877618
Drug: JNJ-38877618: Part 2 — Single ascending dose administered orally in the formulation selected based on Parts 1a, 1b, and 1c (if applicable). The planned dose range for Parts 1 and 2 will be 6 to 1200 mg.
  Arms: JNJ-38877618
Drug: JNJ-38877618: Part 3 — Multiple ascending dose and formulation determined in Part 2 (not to exceed 600 mg) administered orally.
  Arms: JNJ-38877618
Drug: JNJ-38877618: Part 4 (optional) — Single dose and formulation as determined in Part 3 administered orally in older healthy male participant cohort.
  Arms: JNJ-38877618
Drug: Placebo: Parts 1a, 2, 3, and 4 (optional) — Administered orally matched to study drug
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamic effects of single oral doses and multiple oral doses of JNJ-38877618 administered for 7 consecutive days in healthy adult male participants.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), double-blind (individuals and study personnel will not know the identity of study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study in healthy adult male participants aged 18 to 45 years (a single optional cohort in older healthy male participants aged 50 to 65 years may be included). If all optional cohorts are included, up to 144 participants may be enrolled. This study will consist of up to four parts. Part 1 contains up to 3 subparts: Part 1a is a double-blind, placebo-controlled, single ascending dose design (SAD) with a liquid formulation (Formulation A); Part 1b is an open-label (identity of assigned study drug will be known), single dose evaluation of a capsule formulation (Formulation B); and Part 1c is an optional open-label, single dose evaluation of a capsule formulation (Formulation C). Part 2 is the completion of the double-blind, placebo-controlled SAD after a formulation has been selected based on Parts 1a, 1b, and 1c (if applicable). Part 3 is a double-blind, placebo-controlled, multiple ascending dose design (MAD). Doses for Part 3 will be determined based on the safety, tolerability, and pharmacokinetics (study of what the body does to a drug) in Parts 1 and 2. Part 4 is an optional double-blind, placebo-controlled, single dose evaluation in older healthy male participants. Serial pharmacokinetic and pharmacodynamics (study of what a drug does to the body) samples will be collected and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Deemed healthy on the basis of physical examination, medical history, laboratory tests, vital signs, and 12-lead electrocardiogram within protocol-defined parameters performed at screening and Day -1
* Must have good exercise tolerance
* Agrees to protocol-defined use of effective contraception
* Body Mass Index between 20 and 30 kg/m2 and body weight not less than 65 kg
* Non-nicotine user for 6 months prior to screening

Exclusion Criteria:

* Current history of clinically significant medical illness
* History of drug or alcohol abuse within 5 years
* Routine consumption of >450 mg of caffeine per day
* Recent vaccination or acute illness
* Blood donation or major blood loss within 3 months prior to study drug administration
* Use of any prescription or over-the-counter medication (not including paracetamol), or herbal medication within 2 weeks of dosing of the study drug or a proton pump inhibitor within 6 weeks prior to dosing of study drug
* Currently enrolled in an investigational study, or received an investigational drug or vaccine, or used an invasive investigational medical device within 3 months before the planned first dose of study drug
* Plans to father a child while enrolled in this study or within 3 months after the last dose of study drug
* Major surgery within 3 months before or after study participation or minor surgery within 6 weeks before screening, or 30 days after the last study drug administration
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants affected by adverse events by MedDRA system organ class (SOC) and Preferred term (PT) | Up to 30 days after the last dose of study medication
Time to reach the maximum observed plasma concentration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Area under the plasma concentration-time curve from time 0 to 24-hours post dose of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Area under the plasma concentration-time curve from time 0 to infinite time of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Elimination half-life of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
First-order rate constant associated with the terminal portion of the curve of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Total clearance of drug after oral administration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Apparent volume of distribution after oral administration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 4 Day 2)
Maximum observed plasma concentration during a dosing interval at steady state of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Minimum observed plasma concentration during a dosing interval at steady state of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Average plasma concentration over the dosing interval at steady state of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Trough observed plasma concentration at the end of dosing interval of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Time to reach the maximum observed plasma concentration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Area under the plasma concentration-time curve during a dosing interval of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Area under the plasma concentration-time curve during a dosing interval at steady-state of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Total clearance of drug after oral administration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Accumulation index of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)
Apparent volume of distribution at steady-state after oral administration of JNJ-38877618 | Up to 24 hours after last dose of study medication (up to Part 3 Day 8)

SECONDARY OUTCOMES:
Maximum tolerated dose of JNJ-38877618 | Up to 30 days after last dose of study medication (up to Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.
Locations (1):
- Nottingham, United Kingdom